CLINICAL TRIAL: NCT04396860
Title: A Randomized Phase II/III Open-Label Study of Ipilimumab and Nivolumab Versus Temozolomide in Patients With Newly Diagnosed MGMT (Tumor O-6-Methylguanine DNA Methyltransferase) Unmethylated Glioblastoma
Brief Title: Testing the Use of the Immunotherapy Drugs Ipilimumab and Nivolumab Plus Radiation Therapy Compared to the Usual Treatment (Temozolomide and Radiation Therapy) for Newly Diagnosed MGMT Unmethylated Glioblastoma
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-03404; NCI-2020-03404 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-BN007 (Other: NRG Oncology); NRG-BN007 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2020-05-20; First posted 2020-05-21 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-09

CONDITIONS: Gliosarcoma; MGMT-Unmethylated Glioblastoma
MeSH Terms: conditions — Gliosarcoma | interventions — Magnetic Resonance Spectroscopy; Contrast Media; Ipilimumab; CTLA-4 Antigen; Nivolumab; Radiotherapy; Radiation; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (radiation therapy, temozolomide) (Active Comparator): Patients undergo radiation therapy for 5 days per week (Monday-Friday) for a total of 30 fractions over 6 weeks and simultaneously receive temozolomide PO daily for 6 weeks. After radiation, patients may wear the Optune device at the discretion of the patient and their treating physician. Beginning 1 month after radiation therapy, patients receive temozolomide on days 1-5. Treatment repeats every 28 days for up to 12 cycles at the discretion of the treating investigator in the absence of disease progression or unacceptable toxicity. Patients also undergo contrast-enhanced brain MRI throughout the trial.
  Interventions: Procedure: Contrast-enhanced Magnetic Resonance Imaging; Device: NovoTTF-100A Device; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Temozolomide
- Arm II (radiation therapy, ipilimumab, nivolumab) (Experimental): Patients undergo radiation therapy for 5 days per week (Monday-Friday) for a total of 30 fractions over 6 weeks. Starting on the first day of radiation, patients also receive ipilimumab IV over 90 minutes Q4W for 4 doses and nivolumab IV over 30 minutes every 2 weeks until disease progression. Patients also undergo contrast-enhanced brain MRI throughout the trial.
  Interventions: Procedure: Contrast-enhanced Magnetic Resonance Imaging; Biological: Ipilimumab; Biological: Nivolumab; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy

INTERVENTIONS:
Procedure: Contrast-enhanced Magnetic Resonance Imaging — Undergo contrast-enhanced brain MRI
  Other Names: CONTRAST ENHANCED MRI; Contrast-enhanced MRI; MRI With Contrast
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
  Arms: Arm II (radiation therapy, ipilimumab, nivolumab)
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
  Arms: Arm II (radiation therapy, ipilimumab, nivolumab)
Device: NovoTTF-100A Device — Wear Optune device
  Other Names: NovoTTF-100A; NovoTTF-100A System; NovoTTF-100A system (Optune); NovoTTFields; NovoTumor Treatment Fields; Optune; Optune Device
  Arms: Arm I (radiation therapy, temozolomide)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ
  Arms: Arm I (radiation therapy, temozolomide)

SUMMARY:
This phase II/III trial compares the usual treatment with radiation therapy and temozolomide to radiation therapy in combination with immunotherapy with ipilimumab and nivolumab in treating patients with newly diagnosed MGMT unmethylated glioblastoma. Radiation therapy uses high energy photons to kill tumor and shrink tumors. Chemotherapy drugs, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Temozolomide, may not work as well for the treatment of tumors that have the unmethylated MGMT. Immunotherapy with monoclonal antibodies called immune checkpoint inhibitors, such as ipilimumab and nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. It is possible that immune checkpoint inhibitors may work better at time of first diagnosis as opposed to when tumor comes back. Giving radiation therapy with ipilimumab and nivolumab may lengthen the time without brain tumor returning or growing and may extend patients' life compared to usual treatment with radiation therapy and temozolomide.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if adding ipilimumab and nivolumab to radiotherapy significantly prolongs progression-free survival (PFS) versus adding temozolomide to radiotherapy in patients with newly diagnosed glioblastoma (GBM) without MGMT promoter methylation. (Phase II) II. To determine if adding ipilimumab and nivolumab to radiotherapy significantly prolongs overall survival (OS) versus adding temozolomide to radiotherapy in patients with newly diagnosed GBM without MGMT promoter methylation. (Phase III)

SECONDARY OBJECTIVES:

I. To determine if adding ipilimumab and nivolumab to radiotherapy significantly prolongs PFS versus adding temozolomide to radiotherapy in patients with newly diagnosed GBM without MGMT promoter methylation for the phase III part of the study.

II. To determine if adding ipilimumab and nivolumab to radiotherapy significantly increases the 2-year OS rate versus adding temozolomide to radiotherapy in patients with newly diagnosed GBM without MGMT promoter methylation.

III. To evaluate the safety of adding ipilimumab and nivolumab to radiotherapy via comparative frequency between arms of specific adverse events of interest and frequency summaries for all adverse event types.

IV. To evaluate the effect of adding ipilimumab and nivolumab to radiotherapy versus adding temozolomide to radiotherapy on patient reported outcomes (PROs), as measured by the MD Anderson Symptom Inventory - Brain Tumor (MDASI-BT) in patients with newly diagnosed GBM without MGMT promoter methylation.

V. To evaluate the effect of adding ipilimumab and nivolumab to radiotherapy versus adding temozolomide to radiotherapy on selected Patient Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) items in patients with newly diagnosed GBM without MGMT promoter methylation.

VI. To evaluate the impact of adding ipilimumab and nivolumab to radiotherapy versus adding temozolomide to radiotherapy on neurocognitive function (NCF) in patients with newly diagnosed GBM without MGMT promoter methylation.

EXPLORATORY OBJECTIVES:

I. To explore biomarkers in pre-treatment archival tumor tissue that may predict efficacy of ipilimumab and nivolumab as measured by OS, PFS, and 2-year OS rate, such as but not limited to:

Ia. PDL1 expression; Ib. Mutational burden. II. To explore (in the two treatment separately) whether the MGMT protein expression correlates with clinical outcomes including OS, PFS, and 2-year OS rate.

III. To evaluate if MGMT protein expression may be predictive of differential treatment effects between the two treatment arms.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients undergo radiation therapy for 5 days per week (Monday-Friday) for a total of 30 fractions over 6 weeks and simultaneously receive temozolomide orally (PO) daily for 6 weeks. After radiation, patients may wear the Optune device at the discretion of the patient and their treating physician. Beginning 1 month after radiation therapy, patients receive temozolomide on days 1-5. Treatment repeats every 28 days for up to 12 cycles at the discretion of the treating investigator in the absence of disease progression or unacceptable toxicity. Patients also undergo contrast-enhanced brain magnetic resonance imaging (MRI) throughout the trial.

ARM 2: Patients undergo radiation therapy for 5 days per week (Monday-Friday) for a total of 30 fractions over 6 weeks. Starting on the first day of radiation, patients also receive ipilimumab intravenously (IV) over 90 minutes once every 4 weeks (Q4W) for 4 doses and nivolumab IV over 30 minutes every 2 weeks until disease progression. Patients also undergo contrast-enhanced brain MRI throughout the trial.

After completion of study treatment, patients are followed up every 3 months for year 1, then every 4 months for year 2, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* PRIOR TO STEP 1 REGISTRATION:
* No known IDH mutation. (If tested before step 1 registration, patients known to have IDH mutation in the tumor on local or other testing are ineligible and should not be registered)
* Availability of formalin-fixed paraffin-embedded (FFPE) tumor tissue block and hematoxylin & eosin (H&E) stained slide to be sent for central pathology review for confirmation of histology and MGMT promoter methylation status. Note that tissue for central pathology review and central MGMT assessment must be received by the New York University (NYU) Center for Biospecimen Research and Development (CBRD) on or before postoperative calendar day 23. If tissue cannot be received by postoperative calendar day 23, then patients may NOT enroll on this trial as central pathology review will not be complete in time for the patient to start treatment no later than 6 weeks following surgery. Results of central pathology review and central MGMT analysis will generally be conveyed to NRG Oncology within 10 business days of receipt of tissue. Note: In the event of an additional tumor resection(s), tissue must be received within 23 days of the most recent resection and the latest resection must have been performed within 30 days after the initial resection. Surgical resection (partial or complete) is required; a limited biopsy is not allowed because it will not provide sufficient tissue for MGMT analysis

  * Note: The central pathology review and central MGMT results determine eligibility. Therefore, patients may be offered the opportunity to consent REGARDLESS of local pathology and MGMT results, and consent can occur BEFORE local pathology interpretation is finalized and BEFORE local MGMT testing is conducted
* Contrast-enhanced brain MRI within 3 days after surgery

  * MRI with Axial T2 weighted FLAIR {preferred} or T2 turbo spin echo (TSE)/fast spin echo (FSE) and 3-dimensional (3D) contrast-enhanced T1 sequences are required
  * 3D pre contrast-enhanced T1 sequences are strongly suggested
* Women of childbearing potential (WOCBP) and men who are sexually active with WOCBP must be willing to use an adequate method of contraception hormonal or barrier method of birth control; or abstinence during and after treatment
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry
* PRIOR TO STEP 2 REGISTRATION:
* Histopathologically proven diagnosis of glioblastoma (or gliosarcoma as a subtype of glioblastoma) confirmed by central pathology review

  * Note: diagnoses of "Molecular glioblastoma" per the Consortium to Inform Molecular and Practical Approaches to Central Nervous System (CNS) Tumor Taxonomy (c-IMPACT-NOW) criteria or "CNS grade 4" per the World Health Organization (WHO) 2021 criteria are NOT relevant
* MGMT promoter without methylation confirmed by central pathology review. Note: Patients with tissue that is insufficient or inadequate for analysis, fails MGMT testing, or has indeterminate or methylated MGMT promoter are excluded.

  * Note: central pathology review and central MGMT results determine eligibility; local pathology or MGMT results cannot be used for eligibility/randomization
  * Note: patients with methylated MGMT may be considered for enrollment on NRG-BN011
* IDH mutation testing by at least one method (such as immunohistochemistry for IDH1 R132H) must be performed as part of standard of care and no mutation must be found (i.e IDH wildtype). (If a mutation is identified then the patient will be ineligible and must be registered as ineligible at step 2.)

  * Note: this test is not being performed in real time as part of central review and will not be provided to sites from a centrally performed test
* History/physical examination within 28 days prior to step 2 registration
* Karnofsky Performance Status (KPS) >= 70 within 28 days prior to step 2 registration
* Neurologic function assessment within 28 days prior to step 2 registration
* Age >= 18 years
* Hemoglobin >= 10 g/dl (Note: the use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 10.0 g/dl is acceptable) (within 7 days prior to step 2 registration)
* Leukocytes >= 2,000/mm^3 (within 7 days prior to step 2 registration)
* Absolute neutrophil count >= 1,500/mm^3 (within 7 days prior to step 2 registration)
* Platelets >= 100,000/mm^3 (within 7 days prior to step 2 registration)
* Total bilirubin =< 1.5 x institutional/lab upper limit of normal (ULN) (within 7 days prior to step 2 registration)
* Aspartate transaminase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) =< 2.5 x ULN (within 7 days prior to step 2 registration)
* Alanine transferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN (within 7 days prior to step 2 registration)
* Serum creatinine =< 1.5 x ULN OR creatinine clearance (CrCl) >= 50 mL/min (if using the Cockcroft-Gault formula) (within 7 days prior to step 2 registration)
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* For women of childbearing potential (WOCBP), negative serum or urine pregnancy test within 7 days prior to step 2 registration. Note that it may need to be repeated if not also within 3 days prior to treatment start

  * Women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes

Exclusion Criteria:

* Prior therapy for tumor except for resection. For example, prior chemotherapy, immunotherapy, or targeted therapy for GBM or lower grade glioma is disallowed (including but not limited to temozolomide, lomustine, bevacizumab, any viral therapy, ipilimumab or other CTLA-4 antibody, PD-1 antibody, CD-137 agonist, CD40 antibody, PDL-1 or 2 antibody, vaccine therapy, polio or similar viral injection as treatment for the tumor, and/or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways) as is prior Laser interstitial thermal therapy (LITT), Gliadel wafer, radiotherapy, radiosurgery, gamma knife, cyber knife, vaccine or other immunotherapy, brachytherapy, or convection enhanced delivery;

  * Note that 5-aminolevulinic acid (ALA)-mediated fluorescent guided resection (FGR) photodynamic therapy (PDT) or fluorescein administered prior to/during surgery to aid resection is not exclusionary and is not considered a chemotherapy or intracerebral agent
* Current or planned treatment with any other investigational agents for the study cancer
* Definitive clinical or radiologic evidence of metastatic disease outside the brain
* Prior invasive malignancy (except non-melanomatous skin cancer, cervical cancer in situ and melanoma in situ) unless disease free for a minimum of 2 years
* Prior radiotherapy to the head or neck that would result in overlap of radiation therapy fields
* Pregnancy and nursing females due to the potential teratogenic effects and potential risk for adverse events in nursing infants
* History of severe hypersensitivity reaction to any monoclonal antibody
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ipilimumab, nivolumab, or temozolomide
* On any dose of any systemically administered (oral, rectal, intravenous) corticosteroid within 3 days prior to step 2 registration. Inhaled, topical, and ocular corticosteroids are allowed without limitation but must be recorded. Note that treatment with systemically administered corticosteroid after initiating study treatment is allowed as needed
* Patients with known immune impairment who may be unable to respond to anti-CTLA 4 antibody
* History of interstitial lung disease including but not limited to sarcoidosis or pneumonitis
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, defined as New York Heart Association functional classification III/IV (Note: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association functional classification), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, are excluded, as are patients on active immunosuppressive therapy. These include but are not limited to: patients with a history of immune-related neurologic disease, CNS or motor neuropathy, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as autoimmune vasculitis [e.g., Wegener's Granulomatosis]), systemic lupus erythematosus (SLE), connective tissue diseases (e.g., systemic progressive sclerosis), scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome, Hashimoto's thyroiditis, autoimmune hepatitis are excluded because of the risk of recurrence or exacerbation of disease

  * Exceptions: patients with a history of the following conditions are not excluded, unless receiving active immunosuppressive therapy:

    * Vitiligo
    * Type I diabetes
    * Rheumatoid arthritis and other arthropathies
    * Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA)

      * Anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible
* Patients who have evidence of active or acute diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation are also excluded
* Current or planned therapy with warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2026-09-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew B Lassman, Principal Investigator — NRG Oncology
Locations (285):
- United States (285):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - John Muir Medical Center-Concord, Concord, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente-Ontario, Ontario, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Torrance Memorial Medical Center, Torrance, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Lewis Hall Singletary Oncology Center, Thomasville, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - MaineHealth Waldo Hospital, Belfast, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - Maine Medical Partners Neurology, Scarborough, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Good Samaritan University Hospital, West Islip, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Crozer-Keystone Regional Cancer Center at Broomall, Broomall, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Lancaster General Ann B Barshinger Cancer Institute, Lancaster, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Rock Hill Radiation Therapy Center, Rock Hill, South Carolina
  - Avera Cancer Institute at Pierre, Pierre, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Lassman AB, Polley MC, Iwamoto FM, Sloan AE, Wang TJC, Aldape KD, Wefel JS, Gondi V, Gutierrez AN, Manasawala MH, Gilbert MR, Sulman EP, Wolchok JD, Green RM, Neil EC, Lukas RV, Goldlust SA, Snuderl M, Galbraith K, Dignam JJ, Won M, Mehta MP. Dual Immune Check Point Blockade in MGMT-Unmethylated Newly Diagnosed Glioblastoma: NRG Oncology BN007, a Randomized Phase II/III Clinical Trial. J Clin Oncol. 2025 Sep 20;43(27):3032-3040. doi: 10.1200/JCO-25-00618. Epub 2025 Aug 8. PMID 40779733
- [Derived] Woroniecka K, Fecci PE. Immuno-synergy? Neoantigen vaccines and checkpoint blockade in glioblastoma. Neuro Oncol. 2020 Sep 29;22(9):1233-1234. doi: 10.1093/neuonc/noaa170. No abstract available. PMID 32691060

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening required central pathology review confirmation of glioblastoma histology and unmethylated MGMT promotor status in order to proceed to randomization. Of 374 patients registered, 159 patients were randomized.
Period: Overall Study
Arm/Group | Arm I (Radiation Therapy, Temozolomide) | Arm II (Radiation Therapy, Ipilimumab, Nivolumab)
Started | 80 | 79
Randomized | 80 | 79
Adverse Event Population (Randomized, started protocol treatment, and assessed for adverse events) | 74 | 78
Completed (Participants contributing data to results are considered to have completed the study.) | 80 | 79
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Radiation Therapy, Temozolomide) | Arm II (Radiation Therapy, Ipilimumab, Nivolumab) | Total
Number analyzed (Participants) | 80 | 79 | 159
Age, Continuous [Median (Full Range); unit: years] | 59.5 [28 to 77] | 61 [35 to 79] | 60 [28 to 79]
Age, Customized [Count of Participants; unit: Participants]
  ≤ 49 | 15 | 9 | 24
  50 -59 | 25 | 27 | 52
  60 -69 | 30 | 27 | 57
  ≥ 70 | 10 | 16 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 28 | 54
  Male | 54 | 51 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 16
  Not Hispanic or Latino | 73 | 69 | 142
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 71 | 69 | 140
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9
Karnofsky performance status (KPS) [Count of Participants; unit: Participants] — 70 = Cares for self, unable to carry on normal activity or to do active work; 80 = Normal activity with effort, some signs or symptoms of disease; 90 = Able to carry on normal activity, minor signs or symptoms of disease; 100 = Normal no complaints, no evidence of disease.
  Participants
    70 | 10 | 6 | 16
    80 | 24 | 22 | 46
    90 | 37 | 36 | 73
    100 | 9 | 15 | 24
Extent of resection [Count of Participants; unit: Participants]
  Biopsy | 1 | 0 | 1
  Subtotal | 28 | 27 | 55
  Total (gross) | 51 | 52 | 103
Neurologic function [Count of Participants; unit: Participants]
  No symptoms | 22 | 37 | 59
  Minor symptoms | 44 | 27 | 71
  Moderate symptoms (fully active) | 11 | 10 | 21
  Moderate symptoms (required assistance) | 3 | 5 | 8
Recursive partitioning analysis (RPA) class [Count of Participants; unit: Participants] — * Class III: age < 50 and KPS 90-100.
  * Class IV: age < 50 and KPS < 90; OR age ≥ 50 and KPS 70-100 and partially or total resected with no worse than minor neurologic function impairment.
  * Class V: age ≥ 50 and KPS 70-100 and underwent prior partial or total tumor resection with worse than minor neurologic function impairment; OR age ≥ 50 and KPS <70.
  Participants
    III | 9 | 7 | 16
    IV | 58 | 58 | 116
    V | 13 | 14 | 27
Intent to use Optune [Count of Participants; unit: Participants]
  No | 42 | 41 | 83
  Yes | 38 | 38 | 76

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) (Phase II)
Description: Disease progression was confirmed by central review and defined using an adaptation of the Response Assessment in Neuro-Oncology criteria (Wen et al, J Clin Oncol. 2010 Apr 10;28(11):1963-72. doi: 10.1200/JCO.2009.26.3541. Epub 2010 Mar 15) with modification such that the first MRI performed following completion of radiotherapy is the baseline MRI for determination of radiographic disease. Progression-free survival time is defined as time from randomization to the date of first progression, death, or the last progression assessment with no documented progression (censored). Progression-free survival rates were estimated using the Kaplan-Meier method.
Time Frame: From randomization to date of progression, death, or last known follow-up, whichever occurs first. Maximum follow-up time was 19.3 months.
Population: Randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Radiation Therapy, Temozolomide) | Arm II (Radiation Therapy, Ipilimumab, Nivolumab)
Number analyzed (Participants) | 80 | 79
months | 8.5 [7.1 to 10.4] | 7.7 [6.5 to 8.5]
Statistical Analysis 1: Comparison: Arm I (Radiation Therapy, Temozolomide) vs Arm II (Radiation Therapy, Ipilimumab, Nivolumab); For the phase II endpoint, observation of 100 PFS events among the 150 randomized patients (from both arms) provides 95% statistical power to detect an improvement in median PFS from 5.7 months in the control arm to 9.7 months in the experimental arm, corresponding to a hazard reduction of 42% (hazard ratio 0.58) at one-sided significance level of 0.15 (and 87% power for hazard ratio of 0.65 at this same alpha); Test type: Superiority; p = 0.96, Log Rank; Stratified log-rank; Hazard Ratio (HR) = 1.47, 95% CI 2-sided [0.98 to 2.21] — Reference level = Arm 1

2. Primary Outcome: Overall Survival (OS) (Phase III)
Description: Overall survival time is defined as time from randomization to the date of death from any cause or last known follow-up (censored). Overall survival rates were to be estimated by the Kaplan-Meier method.
Time Frame: From randomization to date of death or last known follow-up. Maximum follow-up time was 19.3 months.
Population: Study did not continue to the Phase III component.
Arm/Group | Arm I (Radiation Therapy, Temozolomide) | Arm II (Radiation Therapy, Ipilimumab, Nivolumab)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: PFS for the Entire Cohort (Phase II/III)
Description: as for outcome 1
Time Frame: From randomization to date of progression, death, or last known follow-up. Maximum follow-up time was 19.3 months.
Population: Study did not continue to the Phase III component.
Arm/Group | Arm I (Radiation Therapy, Temozolomide) | Arm II (Radiation Therapy, Ipilimumab, Nivolumab)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Overall Survival at 2 Years
Description: Overall survival time is defined as time from randomization to the date of death from any cause or last known follow-up (censored). Two-year survival rates were to be estimated by the Kaplan-Meier method.
Time Frame: From randomization to two years
Population: Study did not continue to the Phase III component.
Arm/Group | Arm I (Radiation Therapy, Temozolomide) | Arm II (Radiation Therapy, Ipilimumab, Nivolumab)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants by Highest Grade Adverse Event Reported
Description: Common Terminology Criteria for Adverse Events (version 5.0) grades adverse event severity from 1=mild to 5=death. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data.
Time Frame: From randomization to date of last known follow-up. Maximum follow-up time was 19.3 months.
Population: Randomized participants who started protocol treatment and were assessed for adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Radiation Therapy, Temozolomide) | Arm II (Radiation Therapy, Ipilimumab, Nivolumab)
Number analyzed (Participants) | 74 | 78
Participants
  Grade 1 | 6 | 1
  Grade 2 | 19 | 21
  Grade 3 | 38 | 38
  Grade 4 | 9 | 10
  Grade 5 | 0 | 4

6. Secondary Outcome: Change in MD Anderson Symptom Inventory for Brain Tumor (MDASI-BT) at Six Months (Patient Reported Outcomes)
Description: The MD Anderson Symptom Inventory for brain tumor (MDASI-BT) is a 28-item multi-symptom patient-reported outcome measure assessing the severity of symptoms experienced by cancer patients and the interference with daily living caused by these symptoms, with 9 items specific to brain tumors. Each item ranges from 0 (best condition) to 10 (worst condition). A subscale score is the average of the subscale items, given that a specified minimum numbers of items were completed.
Time Frame: Up to 2 years
Reporting Status: Not Posted, anticipated posting 2026-04

7. Secondary Outcome: Neurocognitive Function (NCF)
Time Frame: Up to 2 years
Reporting Status: Not Posted, anticipated posting 2026-04

8. Secondary Outcome: Selected Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) Items
Description: Questions refer to the participants' experiences for the past 7 days of a given symptom in terms of frequency (never, rarely, occasionally, frequently, almost constantly), severity (none, mild, moderate, severe, very severe), interference with usual or daily activities (not at all, a little bit, somewhat, quite a bit, very much).
Time Frame: Up to 2 years
Reporting Status: Not Posted, anticipated posting 2026-04

9. Other Pre Specified Outcome: OS (if the Study Discontinues in Phase II)
Time Frame: At the end of phase II of study
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Tumor Biomarker Analyses
Description: Will assess PD-L1 expression and mutational burden expression specifically.
Time Frame: Up to 4 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: MGMT Protein Expression
Description: Will assess the prognostic value of MGMT protein expression (in terms of predicting clinical outcomes such as PFS, OS, and 2-year OS rate) in the two treatment arms, separately. In addition, will evaluate if MGMT protein expression may be predictive of differential treatment effects between the two treatment arms. Correlation methods and survival modeling will be used to address these questions.
Time Frame: Up to 4 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Randomization to date of last known follow-up. Maximum follow-up time was 19.3 months.
Description: All-cause mortality was assessed in randomized participants. Adverse events were assessed in randomized participants who started protocol treatment and were assessed for adverse events.
Arm/Group | Arm I (Radiation Therapy, Temozolomide) | Arm II (Radiation Therapy, Ipilimumab, Nivolumab)
All-Cause Mortality (participants affected / at risk) | 41/80 | 37/79
Serious Adverse Events (participants affected / at risk) | 29/74 | 45/78
Other Adverse Events (participants affected / at risk) | 70/74 | 70/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Radiation Therapy, Temozolomide) (N=74) | Arm II (Radiation Therapy, Ipilimumab, Nivolumab) (N=78)
Cardiac disorders - Other (Cardiac disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypophysitis (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 4
Colonic perforation (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 4
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Chills (General disorders) | 0 | 1
Disease progression (General disorders) | 0 | 1
Edema limbs (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 1
Fever (General disorders) | 0 | 2
Gait disturbance (General disorders) | 1 | 0
General disorders and administration site conditions - Other (General disorders) | 0 | 1
Autoimmune disorder (Immune system disorders) | 0 | 2
Bone infection (Infections and infestations) | 1 | 0
Encephalitis infection (Infections and infestations) | 0 | 1
Infections and infestations - Other (Infections and infestations) | 0 | 4
Lung infection (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 3
Sinusitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 2 | 0
White blood cell decreased (Investigations) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Dysphasia (Nervous system disorders) | 2 | 1
Edema cerebral (Nervous system disorders) | 3 | 3
Encephalopathy (Nervous system disorders) | 0 | 5
Headache (Nervous system disorders) | 2 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 1
Muscle weakness left-sided (Nervous system disorders) | 1 | 1
Nervous system disorders - Other (Nervous system disorders) | 2 | 2
Paresthesia (Nervous system disorders) | 1 | 2
Seizure (Nervous system disorders) | 5 | 10
Stroke (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Confusion (Psychiatric disorders) | 0 | 3
Delirium (Psychiatric disorders) | 0 | 1
Mania (Psychiatric disorders) | 0 | 1
Bladder perforation (Renal and urinary disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 2 | 6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Radiation Therapy, Temozolomide) (N=74) | Arm II (Radiation Therapy, Ipilimumab, Nivolumab) (N=78)
Anemia (Blood and lymphatic system disorders) | 21 | 26
Sinus tachycardia (Cardiac disorders) | 1 | 4
Tinnitus (Ear and labyrinth disorders) | 4 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 7
Hypothyroidism (Endocrine disorders) | 0 | 9
Blurred vision (Eye disorders) | 8 | 8
Dry eye (Eye disorders) | 1 | 6
Eye disorders - Other (Eye disorders) | 3 | 8
Abdominal pain (Gastrointestinal disorders) | 9 | 7
Colitis (Gastrointestinal disorders) | 0 | 4
Constipation (Gastrointestinal disorders) | 34 | 16
Diarrhea (Gastrointestinal disorders) | 8 | 23
Dry mouth (Gastrointestinal disorders) | 6 | 6
Dysphagia (Gastrointestinal disorders) | 7 | 4
Mucositis oral (Gastrointestinal disorders) | 4 | 5
Nausea (Gastrointestinal disorders) | 32 | 30
Vomiting (Gastrointestinal disorders) | 12 | 16
Chills (General disorders) | 4 | 8
Edema face (General disorders) | 5 | 6
Edema limbs (General disorders) | 12 | 9
Fatigue (General disorders) | 51 | 50
Fever (General disorders) | 2 | 9
Gait disturbance (General disorders) | 9 | 13
Malaise (General disorders) | 1 | 4
Non-cardiac chest pain (General disorders) | 1 | 4
Pain (General disorders) | 6 | 7
Infections and infestations - Other (Infections and infestations) | 8 | 6
Thrush (Infections and infestations) | 5 | 8
Urinary tract infection (Infections and infestations) | 2 | 4
Dermatitis radiation (Injury, poisoning and procedural complications) | 16 | 13
Fall (Injury, poisoning and procedural complications) | 10 | 5
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 4
Alanine aminotransferase increased (Investigations) | 16 | 23
Alkaline phosphatase increased (Investigations) | 5 | 6
Aspartate aminotransferase increased (Investigations) | 9 | 22
Blood bilirubin increased (Investigations) | 10 | 3
Blood lactate dehydrogenase increased (Investigations) | 2 | 4
Creatinine increased (Investigations) | 9 | 8
Investigations - Other (Investigations) | 5 | 4
Lipase increased (Investigations) | 3 | 4
Lymphocyte count decreased (Investigations) | 34 | 18
Neutrophil count decreased (Investigations) | 8 | 9
Platelet count decreased (Investigations) | 24 | 11
Thyroid stimulating hormone increased (Investigations) | 0 | 4
Weight loss (Investigations) | 10 | 18
White blood cell decreased (Investigations) | 14 | 12
Anorexia (Metabolism and nutrition disorders) | 24 | 24
Dehydration (Metabolism and nutrition disorders) | 2 | 8
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 23 | 26
Hyperkalemia (Metabolism and nutrition disorders) | 4 | 0
Hypernatremia (Metabolism and nutrition disorders) | 6 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 | 13
Hypocalcemia (Metabolism and nutrition disorders) | 7 | 7
Hypoglycemia (Metabolism and nutrition disorders) | 6 | 2
Hypokalemia (Metabolism and nutrition disorders) | 9 | 13
Hyponatremia (Metabolism and nutrition disorders) | 13 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 9
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 11 | 18
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 4 | 4
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 5 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 6
Ataxia (Nervous system disorders) | 6 | 0
Cognitive disturbance (Nervous system disorders) | 6 | 4
Concentration impairment (Nervous system disorders) | 0 | 4
Dizziness (Nervous system disorders) | 14 | 17
Dysarthria (Nervous system disorders) | 3 | 4
Dysgeusia (Nervous system disorders) | 10 | 10
Dysphasia (Nervous system disorders) | 13 | 4
Edema cerebral (Nervous system disorders) | 3 | 4
Headache (Nervous system disorders) | 33 | 31
Memory impairment (Nervous system disorders) | 12 | 13
Muscle weakness left-sided (Nervous system disorders) | 8 | 7
Nervous system disorders - Other (Nervous system disorders) | 9 | 5
Seizure (Nervous system disorders) | 15 | 14
Tremor (Nervous system disorders) | 6 | 10
Agitation (Psychiatric disorders) | 4 | 3
Anxiety (Psychiatric disorders) | 6 | 6
Confusion (Psychiatric disorders) | 10 | 13
Depression (Psychiatric disorders) | 5 | 7
Insomnia (Psychiatric disorders) | 19 | 14
Personality change (Psychiatric disorders) | 4 | 0
Urinary frequency (Renal and urinary disorders) | 4 | 1
Urinary incontinence (Renal and urinary disorders) | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 13
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 34 | 29
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 22
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 16
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 8 | 8
Hypertension (Vascular disorders) | 9 | 15
Hypotension (Vascular disorders) | 5 | 5
Thromboembolic event (Vascular disorders) | 7 | 8

LIMITATIONS AND CAVEATS:
This phase II/III trial did not proceed to the phase III component, per the protocol. Therefore, only phase II outcome measures are reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/60/NCT04396860/Prot_SAP_001.pdf
  • Informed Consent Form (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/60/NCT04396860/ICF_002.pdf